CLINICAL TRIAL: NCT07065916
Title: Arm More + Camp: An Implementation Study of a Modified Constraint Induced Movement Therapy Camp for Children With Hemiparesis
Brief Title: Arm More + Camp: An Implementation Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Adam Kirton, Pediatric Neurologist, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REB25-0524
Record Dates: First submitted 2025-06-25; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hemiplegia; Cerebral Palsy Spastic Hemiplegic; Acquired Brain Injury (Including Stroke)
Keywords: Cerebral palsy; Constraint induced movement therapy; Bimanual therapy; Hemiplegia
MeSH Terms: conditions — Hemiplegia; Brain Injuries; Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Constraint Induced Movement Therapy (Other): Constraint Induced Movement Therapy and Bimanual Therapy
  Interventions: Behavioral: Modified Constraint Induced Movement Therapy

INTERVENTIONS:
Behavioral: Modified Constraint Induced Movement Therapy — Constraint Induced Movement Therapy and Bimanual Therapy

SUMMARY:
Our primary aim is to evaluate the implementation cost of a full day modified constraint induced movement therapy camp for children with hemiparesis.

Participants will complete a day camp (9am to 4pm) with constraint induced movement therapy in Week 1 and bimanual therapy in Week 2.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate hemiparesis due to cerebral palsy or acquired brain injury (e.g, traumatic brain injury, stroke)
* Ability to actively extend wrist to neutral and actively flex and extend fingers (at minimum)
* Attend school full-time
* Able to participate in group activities
* Written consent

Exclusion Criteria:

* Severe hemiparesis due to cerebral palsy or acquired brain injury
* No wrist movement on the hemiplegic hand.
* Unable to concentrate for periods of 60-90minutes

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-07-09 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Implementation Cost | From enrolment to the end of outcome data collection at 3 weeks
  Implementation cost covers all resources necessary, including personnel, time, space, and supplies.

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure | Baseline and the end of treatment at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada